CLINICAL TRIAL: NCT00206544
Title: Anti-Estrogens - A Potential Treatment for Bipolar Affective Disorder in Women?
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Alfred (Other)
Collaborators: Stanley Medical Research Institute (Other); National Health and Medical Research Council, Australia (Other)
Responsible Party: Professory Jayashri Kulkarni, Alfred Psychiatry Research Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APRC 77/02; 03T-415; 284319
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2008-10-24 (Estimated); Status verified 2008-10

CONDITIONS: Bipolar Disorder; Mania; Schizoaffective Disorder
Keywords: Bipolar Affective Disorder; Mania; Anti-Estrogen; Schizoaffective Disorder; Mood
MeSH Terms: conditions — Bipolar Disorder; Mania; Psychotic Disorders | interventions — Tamoxifen; Progesterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 1 (Active Comparator): Tamoxifen 40 mg daily
  Interventions: Drug: Tamoxifen
- 2 (Active Comparator): Progesterone 20 mg daily
  Interventions: Drug: Progesterone
- 3 (Placebo Comparator): Placebo daily
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Tamoxifen — 40 mg daily of adjunctive tamoxifen in oral capsule
  Arms: 1
Drug: Progesterone — 20 mg daily of adjunctive progesterone in oral capsule
  Arms: 2
Other: placebo — adjunctive placebo daily in oral capsule
  Arms: 3

SUMMARY:
OBJECTIVE:

To test the use of two adjunctive hormonal agents in a 28 day three-arm, double-blind, placebo-controlled study in the treatment of acute mania/hypomania.

HYPOTHESIS:

That women receiving adjunctive Tamoxifen or Progesterone will demonstrate a more rapid and more substantial decrease in manic symptoms over the course of the study than women receiving adjunctive placebo.

STUDY POPULATION:

Sixty females with a current diagnosis of Bipolar Affective Disorder or Schizoaffective disorder - Manic Phase, according to the operationalised criteria of the Diagnostic and Statistical Manual, 4th edition (DSM-IV) of the American Psychiatric Association.

STUDY MEDICATION:

Tamoxifen. One third of patients (twenty) will be randomized to receive adjunctive Tamoxifen at 40 mg/day for 28 days. The Tamoxifen will be administered within a plain capsule to maintain "blinding" of treatment arm.

Progesterone. One third of patients (twenty) will be randomized to receive adjunctive oral Provera (progesterone) at 20 mg/day. The Progesterone will be administered within a plain capsule identical to that used with Tamoxifen.

Placebo. The remaining one third of patients will be randomized to receive adjunctive placebo (inert substance). The placebo substance will be administered within a plain capsule identical to that used with Tamoxifen and Progesterone.

STUDY EVALUATIONS:

Data will be collected over a 28-day period for each patient. Visits will be performed at baseline, and then at weekly intervals. A total of five visits will be completed for each patient. The following evaluations will be performed:

* Psychiatric evaluation to determine diagnosis. (Baseline visit only)
* General clinical evaluation including medical history, current conditions and a non-invasive physical examination, body weight, vital signs. (Baseline visit only)
* Medication history (baseline and evaluation visits).
* Demographics (baseline visits only).
* Completion of clinical rating scales; CARS-M, PANSS, MADRS, AIMS, Barnes Akathisia scale (BA), and Simpson-Angus scale (SA) (baseline and evaluation visits). A Menstrual Cycle Interview and a cognitive assessment (RBANS) will be performed at baseline and endpoint (day 28) visit.
* Laboratory tests including; Serum levels of mood stabilizer, luteinizing hormone (LH), follicle-stimulating hormone (FSH), Estrogen, Progesterone, Prolactin, dehydroepiandrosterone (DHEA), Testosterone and protein kinase C(PKC) (baseline and evaluation visits).
* Inclusion/exclusion checklist (baseline visit only).
* Informed consent (baseline visit only).

DETAILED DESCRIPTION:
BACKGROUND:

Bipolar Affective Disorder remains an illness with high morbidity and mortality. Mood stabilizers such as lithium and sodium valproate have been described as having their anti-manic effect by targeting protein kinase C (PKC) isozymes (Manji and Lenos, 1999). In rats chronically treated with lithium, there is a reduction of the major PKC substrate MARCKS and a reduction in the hippocampus of the expression of two protein kinase isozymes, alpha and epsilon. Manji et al. (1999) further postulated that PKC inhibitors such as tamoxifen and other estrogen antagonists might represent a novel class of therapeutic agents for the treatment of mania.

Clinical support for the use of "anti-estrogens" in treating mania are found in case reports such as Nelson (1998), and Goldstein (1986), describing the use of danazol in a case of mania, and by Chouinard et al (1987) describing the use of estrogen and progesterone in a case of mania.

A recent preliminary trial by Bebchuk et al, (2000), demonstrated that adjunctive tamoxifen improved in manic symptoms in seven patients. A limitation of their trial was that they failed to standardise the other treatment agents used, which included lithium, antidepressants, anxiolytic and anti-psychotic medications. Mania in women is also noted to have cyclic variations, which is poorly documented and largely anecdotal. This needs further study, and since there is a preponderance of affective disorder in women, we propose conducting a study in women with active symptoms of mania.

OBJECTIVES OF THE STUDY PRIMARY OBJECTIVE To test and compare the use of two adjunctive hormonal agents in a 28 day three-arm double-blind, placebo-controlled study in the treatment of acute mania or hypomania.

SECONDARY OBJECTIVES To examine the impact of hormonal treatments on PKC pathways in women with mania.

To document any observed cyclical variations in the presentation of mania or hypomania in women with bipolar affective disorder and schizoaffective disorder.

ETHICS REVIEW AND INFORMED CONSENT ETHICS APPROVAL The protocol for this study has been approved by the Southern Health Multidisciplinary Ethics Committee and The Alfred Ethics Committee.

INFORMED CONSENT Only patients who are able to give informed consent, (ie. Able to demonstrate an understanding of the objectives of the study and the implications of their role in it), will be recruited into the study. Patients who are extremely psychotic or disturbed will not be approached to enter the study. Involuntary patients who are able to give informed consent will be able to participate and where possible a guardian or relative will be contacted and notified of the patient's involvement. Patients will be advised that their participation is voluntary and that they are free to withdraw from the study at any stage

CONFIDENTIALITY Once a patient agrees to participate in the study, she will be assigned a code number to ensure anonymity. All files will be identified with the patients code number only. Patient's files will be stored in locked filing cabinets with access available to researchers only. Information about the patient will be restricted to the researchers directly involved and the patient's treating doctor.

STUDY POPULATION NUMBERS A target number of 60 patients will be recruited over 3 years. Patients will be recruited from both inpatient and outpatient settings.

WITHDRAWAL CRITERIA

* Patients are free to withdraw from the study at any stage without offering an explanation.
* Patients experiencing any adverse effects which, in the opinion of the investigator, are serious (i.e. life threatening, requiring hospitalisation or medical treatment) will be withdrawn from the study immediately. All patients withdrawn will be followed up until the adverse event has resolved.

STUDY TREATMENTS CONCOMITANT TREATMENTS All patients will participate in standard in-patient and outpatient psychosocial therapies and activities as advised by their treatment team. All patients will receive psychotropic and non-psychotropic medications as per their treatment teams orders. All medications received during the study will be recorded to be included in the analysis.

STUDY MEDICATION Tamoxifen. One third of patients will be randomised to receive adjunctive Tamoxifen at 40mg/day for 28 days. The Tamoxifen will be administered within a plain capsule to maintain "blinding" of the treatment arm.

Progesterone. One third of patients will be randomised to receive adjunctive Provera (progesterone) at 20mg/day. The Progesterone will be administered within a plain capsule identical to that used with Tamoxifen.

Placebo. The remaining one third of patients will be randomised to receive adjunctive placebo (inert substance). The placebo substance will be administered within a plain capsule identical to that used with Tamoxifen and Progesterone.

MEDICATION SIDE EFFECTS Medication side effects are minimised in this study by the short duration of the trial (28 days), the dosing levels used, and by the careful monitoring of side effects at each visit. Possible side effects of Tamoxifen include; hot flushes, nausea, liver enzyme changes, fluid retention, spotting, changes to blood clotting profiles, and light-headedness. Possible side effects of progesterone (medroxyprogesterone acetate) include; nausea, breast tenderness, changes to liver enzymes, blood clotting profile changes, acne and light-headedness.Patients can withdraw consent at any time during the study.

STUDY EVALUATIONS STRUCTURED CLINICAL INTERVIEW FOR DSM-IV (SCID) The structured clinical interview for DSM-III-R (SCID-R Spitzer et al. 1990 see appendix D) will be used to confirm diagnosis for patients entering the study. This will be performed by the treating doctor prior to randomisation. It consists of a structured interview in which the doctor asks set questions regarding symptoms and then rates the reply on a three point scale where 1 = absent or false and 3 = threshold or true.

CLINICIAN ADMINISTERED RATING SCALE FOR MANIA (CARS - M) The CARS-M is a scale devised specifically to measure the symptoms of Mania associated with BPAD. It is administered as a structured clinical interview. The scale comprises of 15 items and assesses the severity of manic and psychotic symptomatology.

POSITIVE AND NEGATIVE SYMPTOM SCHEDULE (PANSS) The PANSS (Kay et al. 1987) will be performed at screening/baseline and at each evaluation visit. The PANSS consists of a Positive Scale (7 positive symptom constructs), a Negative Scale (7 negative symptom constructs) and a General Psychopathology Scale (16 symptom constructs). For each patient, the scale should be administered by the same rater at the same time of day.

MONTGOMERY ASBERG DEPRESSION RATING SCALE (MADRS) The MADRS is a ten item rating scale for rating levels of depression. Each item is rated on a 7-point scale from 0 to 6, where 0 indicates absence of the symptom and 6 indicates extreme presence of the symptom. The time frame for the scale is the previous four weeks.

ABNORMAL INVOLUNTARY MOVEMENT SCALE (AIMS) The AIMS will be completed at screening/baseline and at each evaluation visit. The scale consists of 10 items, each to be rated on a 4-point scale of severity.

SIMPSON-ANGUS SCALE (SAS) The SAS will be completed at screening/baseline and at each evaluation visit. This scale consists of a list of 10 symptoms, each to be rated on a 5-point scale of severity.

BARNES AKATHISIA RATING SCALE The presence and severity of akathisia will be evaluated at baseline and at each follow-up visit on the Barnes Akathisia Rating Scale. The scale consists of four items (objective observation of akathisia by the investigator, subjective feeling of restlessness by the patient, patient distress due to akathisia, and global evaluation of akathisia).

MENSTRUAL CYCLE INTERVIEW To collect information on patient's menstrual history as well as their current menstrual status, a Menstrual Cycle Interview will be administered for pre-menopausal patients. This interview consists of 13 questions related to the patients menstrual cycle and associated issues. The questionnaire can be used in conjunction with serum hormone levels to determine menstrual cycle phase. The questionnaire is administered at baseline and again at the conclusion of the trial. Patients will also be asked to keep a menstrual calendar to register onset and cessation of menstruation.

LABORATORY TESTS

A blood sample will be collected at baseline and at each visit to measure:

1. Serum mood stabiliser levels.
2. PKC activity, using 32P-labelled phosphate transfer techniques and platelets. To be analysed off site at the Mental Health Research Institute.
3. Hormone assays of estrogen, progesterone, luteinising hormone, follicle stimulating hormone and prolactin. These levels give an indication of anti-estrogen activity.

REPEATABLE BATTERY FOR THE ASSESSMENT OF NEUROPSYCHOLOGICAL STATUS (RBANS)

To evaluate cognitive function the RBANS will be administered at baseline and again at the conclusion of the trial. The RBANS comprises 12 subtests that are used to calculate five index scores (Immediate Memory; Visuospatial/Constructional; Language; Attention; and, Delayed Memory) and a total score.

SAFETY ASPECTS ADVERSE EVENTS All adverse events will be recorded by the investigator at each visit. Any adverse events occurring during the course of the study will be followed up once the patient completes the study until such time that the adverse event has resolved.

SCHEDULE OF PATIENT VISITS SCREENING Patients will be screened as soon after admission as possible. After a patient has been deemed eligible to enter the study, informed consent will be obtained. No study procedures will be implemented prior to attainment of informed consent. Where possible, the baseline visit will be completed at the same time as the screening visit.

EVALUATION VISITS A total of five evaluation visits will be performed at baseline, week 1, 2, 3 & 4. All visits will be performed +/- 2 days of the scheduled visit date. At each evaluation visit researchers will check and record adverse events, perform psychopathology rating scales, and collect the blood sample for hormone assay. Participants will be reimbursed $20 per visit to cover the cost of travel.

STUDY MANAGEMENT DATA RECORDING All data gathered will be entered in the patients file under the patients code number. Files will be stored in the research unit in locked filing cabinets. Data entered on computer will be done so using the patients code number for identification. A separate booklet will be used to record data collected at screening, baseline, and evaluation visits. All files will be retained by the hospital for a period of 15 years after completion or discontinuation of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Female patients who have a current diagnosis of Bipolar Affective Disorder (Manic phase) or Schizoaffective Disorder (Bipolar type in manic phase).
* Female patients who are able to give informed consent.

Exclusion Criteria:

* Female patients who are pregnant or lactating.
* Female patients with postpartum psychosis or related disorder.
* Female patients with known abnormalities in the hypothalamo-pituitary gonadal-axis, thyroid dysfunction, central nervous system tumors.
* Female patients taking estrogen preparations such as the oral contraceptive pill.
* Female patients currently taking interacting drugs including warfarin, aminoglutethimide, diuretics, methyldopa, theophylline, fluoxetine, calcium channel blockers and non-steroidal anti-inflammatory drugs.
* Female patients whose psychotic illness is directly due to illicit drugs or who have a history of substance abuse or dependence during the last 6 months.
* Females with any significant unstable medical illness such as cardiovascular disease, renal disease, Addisons disease, thromboembolic disorders, epilepsy, diabetes etc.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2004-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Scores on CARS-M Scale at trial completion | Baseline and weeks 1, 2, 3 and 4

SECONDARY OUTCOMES:
Scores on PANSS at trial completion (4 weeks) | Baseline and weeks 1, 2, 3 and 4
Scores on MADRS at trial completion (4 weeks) | Baseline and weeks 1, 2, 3 and 4
Scores on Adverse Symptom Checklist at trial completion (4 weeks) | Baseline and weeks 1, 2, 3 and 4
Change in hormone levels over trial duration | Baseline and weeks 1, 2, 3 and 4
Scores on RBANS at trial completion (4 weeks) | Baseline and week 4

CONTACTS AND LOCATIONS:
Overall Officials: Jayashri Kulkarni, MBBS, MPM, FRANZCP, PhD, Principal Investigator — Bayside Health / Monash University
Locations (1):
- Bayside Health - The Alfred Hospital, Melbourne, Victoria, Australia

REFERENCES:
- See also: Alfred Psychiatry Research Centre — http://www.med.monash.edu.au/spppm/research/aprc/